CLINICAL TRIAL: NCT01975103
Title: Phase 2 Study of Non-damaging Retinal Laser Therapy Using PASCAL Laser With Endpoint Management Software for Macular Diseases
Brief Title: Non-damaging Retinal Laser Therapy With PASCAL Laser for Macular Diseases
Acronym: EPM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Daniel Lavinsky, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPM-001
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Diabetic Macular Edema; Branch Retinal Vein Occlusion; Chronic Central Serous Retinopathy; Macular Telangiectasia
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: One arm receives laser treatment and second arm received powerless laser treatment as a Sham group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topcon Endpoint management (Experimental): Active laser treatment
  Interventions: Procedure: Topcon Endpoint Management
- Control (Sham Comparator): Powerless (sham) laser treatment
  Interventions: Procedure: Topcon Endpoint Management

INTERVENTIONS:
Procedure: Topcon Endpoint Management

SUMMARY:
This trial seeks to prove the safety and efficacy of photothermal stimulation treatment to diabetic macular edema, chronic central serous retinopathy, macular edema secondary to branch retinal vein occlusion and macular telangiectasia.

DETAILED DESCRIPTION:
Sub-visible, non-damaging photothermal stimulation (532nm) exposures of 100 ms in duration resulted in enhanced expression of heat shock proteins in the retina. To test clinical efficacy of sub-visible retinal therapy using ms-range exposures of visible lasers one needs first to establish proper titration methods necessary to assure on one hand the lack of tissue damage, and on the other hand sufficient hyperthermia to elicit cellular response. We used an algorithm based on computational and experimental data to provide parameters that can cause photothermal stimulation to the retinal pigment epithelium without causing collateral damage to photoreceptors or choroid. This method will be used to treat macular diseases such as diabetic macular edema, branch retinal vein occlusion macular edema, chronic central serous retinopathy and macular telangiectasia.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have macular edema involving the center of the macula with a corresponding leakage on fluorescein angiography.

Thickening of the fovea of at least 300 microns (thickness of the central point in OCT) with a standard deviation of the center point <10% and signal strength of ≥ 5 OCT ILM and borders (internal limiting membrane) and RPE (retinal pigment epithelium) properly identified. Also, the initial OCT must be confirmed by repeated measurements on the same day, with the thickness of the central point being within 10% between measurements. In cases where the OCT imaging program can not properly define the limits of ILM and RPE, if the investigator can obtain an estimate of the thickness of the manual by OCT central point of at least 300 microns, the patient will be considered eligible.

The distance visual acuity in the better eye corrected the study must have an index between 70 and 35 letters inclusive (Snellen equivalent of 20/40 to 20/200).

Clear media and eye pupil dilation adequate to allow fundus photography with good quality.

Intraocular pressure not exceeding 21 mmHg. The ophthalmologist should feel comfortable with the delay of the focal laser treatment (direct and grid, as needed) by at least 12 weeks in the study eye.

Patients with diabetes Type I or Type II as defined by WHO criteria of any gender and age ≥ 18 years.

Ability to provide a written consent. Ability to return for all study visits.

Exclusion Criteria:

* Eyes with scatter photocoagulation (PRP) one month prior the enrollment, or eyes where scatter photocoagulation is required now, or it likely to be needed over the next 6months (for example, eyes with high risk PDR DRS not properly treated with photocoagulation).

Presence of any abnormality that is likely to confound the assessment of the improvement in visual acuity in eyes with macular edema to resolve or improve as an area of hard exudates involving the foveal avascular zone (FAZ - involving 2 or more quadrants centered around the foveal avascular zone), epiretinal membrane associated with signs of contraction and / or significant opacification (ie, striations within the diameter of a disc from the center of the fovea), or the presence of chorioretinal atrophy involving the center of the macula.

Vitreomacular traction determined clinically and / or OCT, which in the opinion of the investigator, contributes to macular edema (associated or cause a detachment of the fovea) and prevents the improvement with treatment.

Atrophy / scar / fibrosis involving the center of the macula, including evidence of atrophy treated with laser within 200 microns of the FAZ.

Patients who received panphotocoagulation, YAG laser, or peripheral retinal cryoablation (for retinal tears) or focal or grid photocoagulation within the last 12 weeks or more of treatment with focal or grid laser.

Significant opacities of the optical medium, including cataracts, which may interfere with visual acuity, assessment of toxicity or photography background. Patients will not be included if they have high probability of requiring cataract surgery within the next year.

Any intraocular surgery within 6 months prior to study entry. Prior peeling of epiretinal membrane or inner limiting membrane. Any major surgical procedure within one month of study entry Prior irradiation of the head region of the eye under study. Any previous pharmacological treatment for DME, BRVO, CSR or MacTel (including corticosteroid intravitreal, subconjunctival or subtenon) or at any time during the last 90 days for any other condition.

Important known allergies to sodium fluorescein dye used in angiography. Acute ocular or periocular infection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 6 months

SECONDARY OUTCOMES:
Central macular thickness on OCT | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lavinsky, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Instituto de Oftalmologia Lavinsky, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Lavinsky D, Sramek C, Wang J, Huie P, Dalal R, Mandel Y, Palanker D. Subvisible retinal laser therapy: titration algorithm and tissue response. Retina. 2014 Jan;34(1):87-97. doi: 10.1097/IAE.0b013e3182993edc. PMID 23873164
- [Derived] Lavinsky D, Silva MOD, Chaves AE, Schneider WFM, Lavinsky F, Palanker D. FUNCTIONAL AND STRUCTURAL EFFECTS OF NONDAMAGING RETINAL LASER THERAPY FOR MACULAR TELANGIECTASIA TYPE 2: A Randomized Sham-Controlled Clinical Trial. Retina. 2021 Mar 1;41(3):487-494. doi: 10.1097/IAE.0000000000002882. PMID 33370517